CLINICAL TRIAL: NCT03158454
Title: Capsula Closure Versus Non-Capsula Closure During Hip Arthroscopy in Danish Patients With Femoroacetabular Impingement (FAI)
Brief Title: Capsula Closure vs. Non-Capsula Closure: Hip Arthroscopy in Danish Patients With Femoroacetabular Impingement (FAI)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Danish EC 1-10-72-279-16
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsula Closure (Other)
  Interventions: Procedure: Capsula Closure
- Non-Capsula Closure (Other)
  Interventions: Procedure: Non-Capsula Closure

INTERVENTIONS:
Procedure: Capsula Closure — The capsular closure is performed with a minimum of two vicryl # 2 resorbable sutures
  Arms: Capsula Closure
Procedure: Non-Capsula Closure — No capsular closure procedure is performed.
  Arms: Non-Capsula Closure

SUMMARY:
The purpose of this study is to investigate whether patients undergoing surgical treatment (hip arthroscopy) of FAI syndrome will positively benefit from capsular closure, in terms of higher scores in validated patient reported outcome measurements, compared to a Group of patients with FAI syndrome where the capsule is left open at the end of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Radiological and symptomatic Femoroacetabular Impingement, where surgery is indicated. Preoperatively a minimum of 3 months of relevant physiotherapeutic treatment should have been performed.

Exclusion Criteria:

* Previous hip surgery in either hip
* Malignant disease
* Recent hip or pelvic fractures
* Arthritic disease
* Hip joint dysplasia
* Legg-Calvé-Perthes
* Slipped Capital Femoris Epiphysis
* Recent (within 6 weeks) medical treatment with corticosteroids
* Language problems of any kind

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported outcome scores (Hagos) | From baseline to 2 year after the operation
  Copenhagen Hip and Groin Outcome Score - Questionnaire - Hip-function Score (0-100)

SECONDARY OUTCOMES:
Change in patient reported outcome scores (Ihot12) | From baseline to 2 year after the operation
  Questionnaire - Hip-function Score (0-100)
Change in patient reported outcome scores (NRS) | From baseline to 2 year after the operation
  Questionnaire - Pain-Score (0-10)
Change in patient reported outcome scores (EQ5D | From baseline to 2 year after the operation
  Questionnaire - health outcome score.
Reoperation | Up to 2 years after surgery
  revision hip arthroscopy/THA/other)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Tage-Hansens Gade 2b, Aarhus, Denmark

REFERENCES:
- [Derived] Mygind-Klavsen B, Kraemer O, Lund B, Krogsgaard M, Holmich P, Lind M, Nielsen TG, Miller LL, Philippon M, Dippmann C. Interportal Capsulotomy Closure Does Not Improve the Results After Hip Arthroscopy at 1-Year Follow-up: A Prospective Randomized Controlled Study. Orthop J Sports Med. 2025 Sep 5;13(9):23259671251363604. doi: 10.1177/23259671251363604. eCollection 2025 Sep. PMID 40917599
- [Derived] Dippmann C, Kraemer O, Lund B, Krogsgaard M, Holmich P, Lind M, Briggs K, Philippon M, Mygind-Klavsen B. Multicentre study on capsular closure versus non-capsular closure during hip arthroscopy in Danish patients with femoroacetabular impingement (FAI): protocol for a randomised controlled trial. BMJ Open. 2018 Feb 10;8(2):e019176. doi: 10.1136/bmjopen-2017-019176. PMID 29440159